CLINICAL TRIAL: NCT06370312
Title: Analysis of Synovial Fluid, Bone and Articular Cartilage From Osteoarthritic First Carpometacarpal Joints in Relationship to Metabolic Risk Factors and Patient-reported Hand Function
Brief Title: Analysis of Articular Biomarkers From Osteoarthritic Thumb Basal Joints
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-07921-01
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis Thumb; Osteoarthritis, Knee; Metabolic Disease
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid from thumb basal joint Bone and cartilage from thumb basal joint Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Trapeziectomy — Patients scheduled for trapeziectomy due to thumb basal joint osteoarthritis are invited to participate. Synovial fluid is aspirated before the joint is opened. Bone and cartilage are collected. Blood samples are obtained preop. Patients are measured with grip strength, pinch strength, range of thumb motion, body mass index, central obesity and blood pressure.

SUMMARY:
The study project aims at examining molecular markers in synovial fluid, bone and articular cartilage from osteoarthritic thumb basal joints. The degradation of extracellular matrix (ECM) proteins in thumb basal joints will be evaluated in association to the metabolic profile of the patient, but we also aim to compare the ECM degradation and inflammatory profiles with articular cartilage degradation ECM profile from knee joints with osteoarthritis. A third aim is to evaluate associations between patient-reported hand function, pain, strength and range of thumb motion to analyses of synovial fluid.

DETAILED DESCRIPTION:
Patients scheduled for trapeziectomy on the basis of thumb basal joint osteoarthritis will be asked to participate. Synovial fluid from the thumb basal joint is aspirated before the joint is opened. The trapezium bone and cartilage is harvested. Blood samples to evaluated lipid profile and glucose intolerance is drawn. Blood pressure and measurements of obesity is taken. Patients are also examined at baseline and 1 year postop with grip strength, pinch strength, range of thumb motion and asked to fill in patient-rated outcome measures; QuickDASH and NRS pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 25 years
* Radiologically confirmed and symptomatic thumb basal joint osteoarthritis (OA) planned for trapeziectomy

Exclusion Criteria:

* Previous surgery to the affected thumb basal joint
* Post-traumatic thumb basal joint OA
* Rheumatoid arthritis or other chronic inflammatory arthritis, history of psoriasis affecting joints, gout or pseudogout
* Ongoing infection in the hand or wrist
* Inability to co-operate with the follow-up protocol or to assimilate information about the study protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction)
* Systemic or intra-articular glucocorticoids or intraarticular platelet-rich plasma or hyaluronic acid injections in the affected joint within 3 months prior to enrollment

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients fulfilling the eligibility criteria and are scheduled for surgery at any of two study centres; Department of hand surgery, Skane university hospital or Aleris Malmö Arena (private clinic), due to symptomatic thumb basal joint OA are invited to participate. Indications for surgery at these to clinics are; 1) persistent pain and pain at rest, 2) have tried conservative treatment with inadequate effect.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum cholesterol levels | Serum cholesterol levels are drawn at baseline (i.e. the day of surgery)
  Blood samples are drawn from the patients and analysed according to Swedish laboratory standards

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Brogren, MD, PhD, Principal Investigator — Department of hand surgery, Region Skåne
Locations (2):
- Sweden (2):
  - Department of Hand Surgery, Skane University Hospital, Malmo, Skåne County
  - Aleris Specialistläkare Hyllie, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No
No sharing